CLINICAL TRIAL: NCT00496184
Title: Topical Application of Nifedipine Cream for the Treatment of Vulvar Vestibulitis Syndrome
Brief Title: Efficacy Study of Topical Application of Nifedipine Cream to Treat Vulvar Vestibulitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20050989
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2008-05-08 (Estimated); Status verified 2008-05

CONDITIONS: Vulvar Diseases; Vulvar Pain; Vestibulitis; Vestibulodynia; Vulvodynia
Keywords: Nifedipine treatment; Vestibulitis; Placebo
MeSH Terms: conditions — Vulvar Diseases; Vulvodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Nifedipine cream topical application

SUMMARY:
To evaluate the use of topical application of Nifedipine cream for the treatment of Provoked localized Vulvodynia (vestibulitis, vestibulodynia).

DETAILED DESCRIPTION:
30 women aged 18-45 diagnosed with Provoked localized Vulvodynia will be included. 10 women will use topical Nifedipine cream 0.2% 4 times a day for 6 weeks (except for menstrual period). 10 other women will use topical Nifedipine cream 0.4% 4 times a day for 6 weeks (except for menstrual period).

10 women will be a control group and will use a placebo cream. The study will be randomized and double blind. Participants will be examined before starting the treatment, at the end of the treatment and 3 months after completion the treatment. A special detailed questionnaire has been prepared in three languages and will be used to compare dyspareunia and associate variables between the groups.

The Q-tip tests will be performed and findings will be drawn in each examination. Differences between the groups will be examined, and uni- and multi-variate analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Women diagnosed with vestibulitis according to Friedrich's criteria:

   * Severe pain with vestibular touch or attempted vaginal entry.
   * A positive Q-tip test: pain produced by touching the vestibule with a cotton tipped applicator.
   * Physical findings limited to varying degree of vestibular erythema.
2. Non-pregnant women aged 18-45.
3. Women use effective contraception and are not interested in becoming pregnant during the study period.
4. No known Nifedipine allergy.
5. No medical diseases.

Exclusion Criteria:

1. Women who have undergone vestibulectomy.
2. Active vaginal or pelvic infection.
3. A medical disease uch as Diabetes, immune suppression.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Complete resolution of vestibulitis. | Participants will be examined before starting the treatment, at the end of the treatment and 3 months after completion the treatment, using the questionnaire and the Q-tip applicator for detection of vestibular sensitivity.

SECONDARY OUTCOMES:
Safety of the Nifedipine treatment. | Participants will be examined before starting the treatment, at the end of the treatment and 3 months after completion the treatment, using the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Bornstein, MD, Principal Investigator — Western Galilee Hospital, Nahariya, Israel; Doron Zarfati, MD, Principal Investigator — Western Galilee Hospital, Nahariya, Israel
Locations (2):
- Israel (2):
  - Colposcopy Clinic, Obstetrics and Gynecology Department, Western galilee Hospital, Nahariya
  - Department of Obstetrics and Gynecology, Nahariya

REFERENCES:
- [Background] Walsh KE, Berman JR, Berman LA, Vierregger K. Safety and efficacy of topical nitroglycerin for treatment of vulvar pain in women with vulvodynia: a pilot study. J Gend Specif Med. 2002 Jul-Aug;5(4):21-7. PMID 12192883
- [Background] Nelson R. Non surgical therapy for anal fissure. Cochrane Database Syst Rev. 2003;(4):CD003431. doi: 10.1002/14651858.CD003431. PMID 14583976
- [Background] Bornstein J, Zarfati D, Goldik Z, Abramovici H. Vulvar vestibulitis: physical or psychosexual problem? Obstet Gynecol. 1999 May;93(5 Pt 2):876-80. doi: 10.1016/s0029-7844(98)00535-3. PMID 10912437